CLINICAL TRIAL: NCT03298776
Title: I-Scan a Novel Endoscopic Tool for the Macroscopic Identification of Mucosal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STH18011
Record Dates: First submitted 2017-09-18; First posted 2017-10-02 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard white light endoscopy (Active Comparator): Patients will undergo the standard of care which is standard white light endoscopy
  Interventions: Diagnostic Test: Standard endoscopy
- Endoscopy and I-Scan (Experimental): Patients will undergo standard of care endoscopy plus the I-Scan
  Interventions: Device: I-Scan

INTERVENTIONS:
Device: I-Scan — I-Scan is a digital enhancement technique. These endoscopes already have greater definition compared to many standard endoscopes but they also utilise a 'zoom' function and digital image enhancement.
  Arms: Endoscopy and I-Scan
Diagnostic Test: Standard endoscopy — Patients referred for standard endoscopy to receive standard of care only
  Arms: standard white light endoscopy

SUMMARY:
The use of endoscopy for the diagnosis of gastrointestinal diseases has continued to increase in recent years.

Endoscopy provides an advantage over other noninvasive or minimally invasive procedures in that it allows both direct visualisation of the mucosa but direct and accurate sampling of abnormalities for histological examination. However standard endoscopy does have some limitations particularly with small lesions and pan mucosal changes. Some lesions may be entirely benign and require no further intervention but as a result of difficulty with accurate endoscopic characterization of lesions in many cases unnecessary biopsies or polypectomies are undertaken. Therefore any technology that can augment the use of standard endoscopy to minimise unnecessary intervention should be encouraged. IScan is a digital enhancement technique available with Pentax endoscopes. There have been other novel endoscopic advances for example, Narrow band imaging but these have not been adopted widely for a number of reasons including technical difficulties or patient tolerability. The aim of this study is to assess whether Pentax IScan technology is a reliable method of improving our recognition of macroscopic mucosal lesions compared to standard white light endoscopy

DETAILED DESCRIPTION:
All patients recruited will undergo standard endoscopy using current generation Pentax endoscopes. These endoscopes are widely used for standard endoscopic procedures. All of the endoscopes that will be used have the I-scan function which is controlled by the operator. Therefore there will be no difference between the groups randomised to I-Scan or standard endoscopy, other than a very slight difference in duration for I-scan, which the patient is unlikely to detect. We have received no funding from Pentax for the use of their endoscopes.

Following recruitment patients will be randomly allocated to receive standard white light endoscopy or standard white light endoscopy plus I-Scan using a random number generator at www.random.org with possible values of 0 or 1. Those with a 0 will receive standard endoscopy and those with a 1 will receive standard endoscopy plus I-Scan. Both arms will undergo standard endoscopic evaluation including appropriate biopsies by fully trained experienced endoscopists with Joint Advisory Group (JAG) accreditation for endoscopy. The investigators will be initially blinded to the indication for endoscopy until the I-Scan has been utilised at which point the indication will be revealed to ensure patient safety. Patients will have biopsies only by the clinical indication. No extra biopsies that would not normally be clinically justified will be taken. Following the procedure all patients will be asked to evaluate the tolerability of their test using a validated 10 point likert scale. All procedures will be recorded on an anonymised basis using a unique research identifier and subsequently reviewed by other expert endoscopists within the department to allow us to accurately assess the reliability and interobserver variability of the test. Each of the endoscopists will be fully trained in standard endoscopy and will be blinded to the indication for the procedure.

The study will be a randomised controlled trial. Given the nature of the study it is not possible to blind the investigators to the procedure type. The investigator carrying out the procedure will however be blinded to the indication for the procedure until the I-Scan has been used as this could lead to bias. The endoscopists reviewing the images will be blinded to all patient information and indications for the endoscopy throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending for a routine diagnostic endoscopic procedure where Pentax endoscopes are in use at the endoscopy unit at the Royal Hallamshire Hospital.

Exclusion Criteria:

* Patients attending for a therapeutic endoscopic procedure.
* Patients with a known endoscopic diagnosis
* Patients with abnormal coagulation or any other contraindication to use of standard biopsy or polypectomy techniques used in routine diagnostic endoscopic procedures
* Patients who are unable to understand English or give informed consent
* Patients under the age of 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Clarity of mucosal lesions found using I-Scan | through study completion, on average one year
  The endoscopic assessment of mucosal lesions using standard endoscopy and standard endoscopy plus I-Scan Will be compared to histological assessment where this is indicated. Interobserver variability of assessment of mucosal lesions will be compared between endoscopic techniques

SECONDARY OUTCOMES:
Patient reported tolerability of I-scan procedure | through study completion, on average one year
  The use of the I-scan results in a slight prolongation of the endoscopy procedure. A ten point likert patient reported questionnaire will assess patient tolerability of the I-scan

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD